CLINICAL TRIAL: NCT00499538
Title: A Single Dose Bioavailability Study of 3 New Formulations of SKI-606 (500 mg) Compared With a Reference Capsule and an Oral Solution in Healthy Adult Subjects
Brief Title: Study Evaluating 3 New Formulations of SKI-606 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 3160A4-1109
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
Keywords: healthy subjects
MeSH Terms: interventions — bosutinib

INTERVENTIONS:
Drug: SKI-606

SUMMARY:
To evaluate the comparative bioavailability of 3 new tablet formulations of SKI-606 with a reference capsule and an oral solution in healthy subjects.

ELIGIBILITY:
Criteria:

* Healthy male and female aged 18 to 50 years.
* Women of nonchildbearing potential (WONCBP).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-07; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The data from this study along with in vitro data will be used to explore in vitro/in vivo correlation for SKI-606 to support formulation development.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- San Antonio, Texas, United States